CLINICAL TRIAL: NCT00467493
Title: A Partial Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Anastrozole, an Aromatase Inhibitor, on Endometrial Thickness in Healthy Premenopausal Women When Dosed at Various Times During the Menstrual Cycle (Protocol M-001)
Brief Title: Partial Double-Blind, Placebo-Controlled Study to Assess the Effect of Anastrozole on the Endometrium in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meditrina Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-001
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Menstruation Disorders
MeSH Terms: conditions — Menstruation Disturbances | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Anastrozole - A (Experimental): Treatment for 26 consecutive days
  Interventions: Drug: Anastrozole
- Anastrozole -B (Experimental): Treatment for 7 consecutive days early in menstrual cycle
  Interventions: Drug: Anastrozole
- Anastrozoe - C (Experimental): Treatment for 7 consecutive days mid follicular phase
  Interventions: Drug: Anastrozole
- Anastrozole - D (Experimental): Treatment for 7 consecutive days - mid cycle
  Interventions: Drug: Anastrozole
- Anastrozole - E (Experimental): Treatment for 7 consecutive days - luteal
  Interventions: Drug: Anastrozole
- Anastrozole - F (Placebo Comparator): Treatment with placebo for 26 consecutive days
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole

SUMMARY:
Aromatase inhibitors have been approved for use in postmenopausal women to treat and prevent breast cancer. They act by blocking the action of the enzyme, aromatase, that is necessary for the production of estradiol. This class of drugs, aromatase inhibitors, are very effective in reducing estradiol levels in postmenopausal women and in treating estrogen receptor positive breast cancers. This study is examining the effect of a specific inhibitor, anastrozole, on endometrial thickness in premenopausal women. The endometrium is sensitive to estradiol and also has local aromatase which, if inhibited, may result in reduced endometrial thickness. The main hypothesis is that anastrozole can be administered at any time during the menstrual cycle and reduce endometrial thickness compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 25 and 45 and pre-menopausal;
* Non-lactating and not pregnant
* able to follow the schedule of procedures
* able to freely provide informed consent
* have clinically acceptable physical examination and safety laboratory studies

Exclusion Criteria:

* current use of any form of systemic contraceptive
* have self-reported irregular menstrual cycles
* intercurrent illness(es) detected on the screening physical
* unwilling or unable to use barrier methods of contraception
* have evidence of endometrial polyps or myomata on TVU/SIS that would interfere with endometrial thickness measurement
* detection of ovarian cyst(s) during adnexal examination on screening TVU/SIS measuring greater than 5 cm
* have history of, or current cancer, on any form exclusive of basal cell carcinoma
* BMI >= 35
* history of alcohol or drug abuse in the past 5 years
* unwilling or unable to undergo study procedures within the necessary time frames
* history or current liver abnormalities as defined by ALT or AST > 2X ULN
* treated or untreated diabetes defined as fasting blood sugar >= 126 mg/dL
* untreated hypertension
* impaired renal function by estimated creatinine clearance < 80mL/min
* have estradiol levels < 20 pg/ml and FSH levels > 40 mIU/mL or
* have a history of adverse reaction any aromatase inhibitor

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2007-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness as measured by transvaginal ultrasound, safety | Over one menstrual cycle

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jasper Research Clinic, Kalamazoo, Michigan
  - University Women's Care, Southfield, Michigan